CLINICAL TRIAL: NCT07346846
Title: A Phase 1 First-in-human Study of BGM-2121 in Patients With Advanced Solid Tumors
Brief Title: A Study of BGM-2121 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioGate Precision Medicine Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGM-2121-001
Record Dates: First submitted 2025-11-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BGM-2121 (Experimental)
  Interventions: Drug: BGM-2121

INTERVENTIONS:
Drug: BGM-2121 — BGM-2121 treatment

SUMMARY:
This study is to explore the safety, tolerability, pharmacokinetics, and preliminary efficacy of BGM-2121 in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged ≥ 18 years,
2. Has a confirmed diagnosis of advanced solid tumor(s),
3. The subject has received and failed standard-of-care anti-cancer therapy
4. Has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST)
5. ...

Exclusion Criteria:

1. Has any ongoing toxicity from previous anti-cancer treatments
2. Has signs or symptoms of end-stage organ failure, major chronic illnesses other than cancer(s)
3. History of another primary malignancy within the last three years
4. ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | From first dose through the DLT evaluation period (28 days)
  Number and type of DLTs observed following administration of BGM-2121 at different dose levels, assessed according to protocol-defined criteria.
Treatment Discontinuation Due to Drug-Related Adverse Events | From first dose through study completion, an average of 1 year
  Number of participants who permanently discontinue BGM-2121 due to drug-related adverse events, graded per CTCAE v5.0.
Incidence of Treatment-Emergent and Treatment-Related Adverse Events | From first dose through 6 weeks after the last dose of study treatment
  Incidence, type, and timing of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs), graded per CTCAE v5.0.
Number of Participants With Grade ≥3 Laboratory Abnormalities | From first dose through study completion, an average of 1 year
  Number of participants experiencing Grade 3 or higher laboratory abnormalities, including hematology and serum chemistry parameters, based on CTCAE v5.0 criteria
Changes in Electrocardiogram (ECG) Parameters | From baseline through study completion, an average of 1 year
  Change from baseline in ECG parameters, including QT/QTc interval, PR interval, and QRS duration.

SECONDARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) to establish RP2D | From first dose through the DLT evaluation period (28 days)
  MTD of BGM-2121 in subjects with advanced solid tumors, used to determine the recommended Phase 2 dose (RP2D).
Incidence of Anti-Drug Antibodies (ADAs) | From first dose through 6 weeks after the last dose of study treatment
  Percentage of subjects who develop treatment-emergent ADAs during the study.
Peak Serum Concentration (Cmax) of BGM-2121 | From first dose through 30 days after the last dose
  Cmax derived from serum concentration data.
Area under Curve (AUC) of BGM-2121 | From first dose through 30 days after the last dose
  AUC derived from serum concentration data.
Objective Response Rate (ORR) | From baseline through study completion, an average of 1 year
  Percentage of subjects with complete or partial response according to RECIST 1.1 criteria.
Progression-Free Survival (PFS) | From first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 80 weeks
  Time from first treatment to documented disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No